CLINICAL TRIAL: NCT03011086
Title: Evaluation of Auto Antibodies in Oral Sub Mucous Fibrosis - a Clinico-pathological Study
Brief Title: Evaluation of Auto Antibodies in Oral Sub Mucous Fibrosis
Status: Completed | Type: Observational
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, NALLAN CHAITANYA, ASSOCIATE PROFESSOR, DEPARTMENT OF ORAL MEDICINE AND RADIOLOGY, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Other Study IDs: PMVIDS/OMR/0016/2014
Record Dates: First submitted 2016-11-07; First posted 2017-01-05 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Oral Submucous Fibrosis
Keywords: Autoantibodies, Oral Submucous Fibrosis
MeSH Terms: conditions — Oral Submucous Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- oral sub mucous fibrosis: patients suffering with oral sub mucous fibrosis due to gutka/pan chewing confirmed by clinical examination
- control group: patients having gutka/ pan chewing habit without oral sub mucous fibrosis in oral cavity

SUMMARY:
The etiology of OSMF is considered to be multifactorial. However, Role of autoimmunity had been suggested as one of the factors but remains unproven.

The present study is undertaken to evaluate the presence of auto antibodies in OSMF patients to pave a way for new arena of treatment with the etiology of this persistent condition

DETAILED DESCRIPTION:
Oral submucous fibrosis (OSMF) is a potentially malignant disorder affecting any part of the oral cavity, sometimes pharynx associated with juxta epithelial fibrosis causing progressive trismus leading to dysphagia. It is mainly seen in the Asian countries with more prevalence in India.

Etiology of OSMF is considered to be multifactorial. However, it is strongly associated with the use of arecanut in various forms and also in combination with other compounding factors. Autoimmunity had been suggested as one of the factors yet unproven.

Few studies reveal that there is high incidence of Autoantibodies including antinuclear (ANA), Anti smooth muscle (SMA), Anti thyroid microsomal (TMA), and anti reticulin antibodies in OSMF patients. These findings have not been consistent in further studies which needs further more research in this.

A study concentrated on quantitation of circulating immune complexes (CIC) levels which was established in patients with oral cancer and oral precancerous lesions. The levels were compared with that in normal controls and chronic chewers of betel quid with no signs of any disease. Both patients with oral cancer and oral precancerous lesions had elevated CIC when compared to both the control groups. The most interesting observations were (a) the CIC levels in the chewing controls were significantly raised when compared to normal controls; and (b) the CIC levels in the patients with premalignant lesions were elevated almost to the same levels as in the oral cancer patients.

HLA-typing was carried on areca nut chewers. however, it was unable to demonstrate a specific pattern of HLA-antigen frequencies in chewers with or without the disease. It is not necessarily a HLA-associated susceptibility in Oral Submucous Fibrosis.

Due to less number of articles published on autoantibodies, this study is done to evaluate the presence of such auto antibodies in OSMF patients thereby paving way for new arena of treatment on par with the etiology of this persistent condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing for the study.
* A positive history of chewing arecanut, and/or smoking tobacco and alcohol.
* Patients with clinical and histopathological features of oral submucous fibrosis.
* Patients with OSMF not under any treatment for the same

Exclusion Criteria:

* Unwilling patients who do not want to be part of the study.
* Patients with known autoimmune disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total number of patients were 70 patients (Group A- 35 OSMF patients, Group B- 35 controls) of both the genders
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of auto antibodies in oral sub mucous fibrosis | one and half year
  The subjects in the study suffering from oral submucous fibrosis will be clinically evaluated and graded based on criteria given by Khanna et al classification. All the subjects included in the study will also be subjected to serum analysis for presence of auto antibodies in their serum by Titerplane technique.

CONTACTS AND LOCATIONS:
Overall Officials: NALLAN CHAITANYA, MDS, Principal Investigator — ASSOCIATE PROFESSOR
Locations (1):
- Panineeya Institute of Dental Sciences, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No